CLINICAL TRIAL: NCT06583629
Title: Effect of Emotion Freedom Technique on Perceived Stress, Resilience and Sexual Satisfaction Among Women After Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Alaa El Din Moustafa Hamed Abd Elaleem, Lecturer of Psychiatric and Mental health Nursing, Helwan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: FMBSUREC/03122023/ Mohamed
Record Dates: First submitted 2024-08-28; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Stress; Sexual Satisfaction; Mastectomy
Keywords: Emotional Freedom Technique; Stress; Resilience; Sexual satisfaction
MeSH Terms: conditions — Orgasm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enrolled participants (Experimental)
  Interventions: Behavioral: Emotional Freedom Technique

INTERVENTIONS:
Behavioral: Emotional Freedom Technique — EFT is a self-help technique that incorporates conscious awareness of thoughts and feelings with a gentle touch involving tapping with fingertips on acupuncture/acupressure points on the face, hands, and body. EFT also helps relieve primary physical and emotional symptoms. Gary Craig created EFT, which involved lightly tapping on the body on 12 acupressure sites (also known as acupoints). This acupoints are situated along the body's meridians, or virtual energy channels
  Other Names: Tapping

SUMMARY:
A quasi-experimental design was utilized, involving a convenient sample of 112 Egyptian mastectomized women. Data were collected and analyzed to determine the correlations between the variables of interest.

DETAILED DESCRIPTION:
Aim of the Study:

This study set out to evaluate the effect of emotion freedom technique on perceived stress, Resilience and sexual satisfaction among women after mastectomy.

Setting and study design:

The study was conducted in the surgical department, Beni-Suef University Hospital, at Beni-Suef Governorate, Egypt. A quasi-experimental design was utilized to carry out the study.

Participants:

A total of 112 Egyptian women who had undergone mastectomy were recruited based on the following inclusion criteria: a) absence of any psychiatric diagnoses, b) no prior exposure to courses on emotional freedom techniques, c) no chronic illnesses, and d) willingness to participate in the study.

Study instruments and measures:

For this study, a well-structured interview using a previously prepared questionnaire with the participants using the participants' mother tongue (Arabic) was employed. The researchers developed the questionnaire, incorporating relevant Connor-Davidson Resilience scale items, Perceived Stress Scale, and the Sexual Satisfaction Index from related studies. The instruments were translated from English to Arabic at the Center for Specialized Languages, Faculty of Arts, Helwan University. A panel of experts in psychology, psychiatry and psychiatric nursing then evaluated the instrument's validity and suitability for use with mastectomized women. The questionnaire's validity was further confirmed through a pilot study involving 10 participants. Then the questionnaire was distributed by the researchers through performing an interview with the participants in the surgical department, Beni-Suef University Hospital.

This research instrument encompasses four primary sections, the first one containing the participant's basic and educational information, including items such as: age, educational level, place of residence, marital status, occupation, economic status and medical history of the women. The second section was Connor-Davidson Resilience Scale (CD-RISC) which was developed Kathryn and Jonathan, (2003). Connor-Davidson Resilience Scale (CD-RISC) comprises 25 items that measure resilience or capacity to change and cope with adversity. Respondents indicated their response on a 5-point Likert scale with higher scores indicating greater resilience. Scoring criteria: As for the scoring system of the CD-RISC contains 25 items, all of which carry a 5-point range of responses, as follows: not true at all (0), rarely true (1), sometimes true (2), often true (3), and true nearly all of the time (4). The scale is rated based on how the subject has felt over the past month. The total score ranges from 0-100, with higher scores reflecting greater resilience. Cronbach's alpha coefficient for the full scale was 0.89.

The third research instrument's part was the Perceived Stress Scale (PSS-10) which was developed by Cohen and colleagues, (1983). The Perceived Stress Scale (PSS) is widely considered the gold standard instrument for measuring stress perception. This questionnaire is used to assess the degree to which a respondent finds circumstances in their life to be unpredictable, uncontrollable, and/or overwhelming. Questions on the PSS ask the respondent to rate their feelings and thoughts for the past month indicating that a relatively recent time frame is assessed. PSS designed to measure the degree to which situations in one's life are appraised as stressful. This version of the PPS had 10 items: four positive items (items 4, 5, 7, 8) and six negative items (items 1, 2, 3, 6, 9 and 10). Each item is scored on a 5-point scale, ranging from 0 (never) to 4 (very often). The positive elements' ratings are reversed, for example, 0=4, 1=3, 2=2, etc., and then summing across all 10 items, a higher score indicates more perceived stress. We evaluated the internal consistency of the questionnaire with Cronbach's alpha, resulting in a satisfactory value of 0.82.

The fourth part of the research instrument was the Sexual Satisfaction Index (SSI) which was developed by Leth-Nissen and colleagues, (2021). There were nine items in this edition of the SSI: five positive items (items 1, 2, 3, 8, and 9) and four negative ones (items 4, 5, 6, and 7). Every item is scored on a 5-point rating system, with the negative ratings being reversed and ranging from 1 (strongly disagree) to 5 (strongly agree). The SSI's total score falls between 1 and 45. A greater level of sexual satisfaction is indicated by a higher sum score. Estimates of internal reliability for the SSI produced acceptable Cronbach's alpha coefficients to the full scale 0.88.

Procedures:

The data collection for this study was instituted after obtaining the ethical approval from the faculty of medicine at Beni-Suef University, followed by the approval from the hospital authorities to conduct the current study after an explanation of the aim of the study.

The researchers prepared the research instruments after reviewing related articles and periodicals. The instrument was translated from English to the participant's mother tongue, "Arabic," at the Center for Specialized Languages of the Faculty of Arts, Helwan University. A panel of experts in psychology, psychiatry, and psychiatric/mental health nursing then evaluated the instrument's validity and suitability for use with nursing students.

The survey was successfully conducted with participants in the hospital in the form of a well-structured interview, where the researchers met the participants, explained the aim of the study to them, assessed their ability to participate, and obtained their written informed consent; the informed consent, explaining the study's aim, confidentiality guarantees, and the ability to withdraw from the study at any time without any fear. Then the data was collected. The emotional freedom technique was applied through various phases. The preparatory phase involved reviewing the studies and available literature related to the research problem and theoretical knowledge using evidence-based articles, textbooks, internet periodicals, and journals. The assessment phase, in which the researchers communicated with the accountable nursing supervisors in the surgical department daily to find out how many patients were recently admitted to the surgical department and if they fulfilled the inclusion criteria. The researchers clarified the nature and the aim of the study to all participants who were involved in the study after taking their written approval of participation. The researchers interviewed the participants (pre-the emotional freedom technique interventions) to complete the socio-demographic, perceived stress, resilience, and sexual satisfaction. The interview lasted between 25 and 35 minutes.

Planning Phase (Development of Emotional Freedom Technique Interventions): The objectives were formulated with careful consideration of the needs of the women involved, drawing on recent significant research and expert validation from the nursing field. These objectives were revised and refined based on expert feedback to ensure they could be applied in various ways. One such approach included the creation of a booklet, which highlighted the key aspects of the emotional freedom technique specifically for women who had undergone mastectomies. The booklet, designed by researchers, was written in simple Arabic and accompanied by illustrative photos. Implementation phase: The implementation of emotional freedom technique interventions was carried out by the researchers. Interventions were provided three times per week. The emotional freedom technique, with approximately (55 minutes) included theoretical information about breast cancer, signs and symptoms, treatment and its effect on stress, resilience, and sexual satisfaction (25 minutes), and steps of applying the emotional freedom technique (30 minutes). The evaluation phase aimed to reevaluate the participants to find any variations in their baseline response level following the intervention phase. Both before and after using the emotional freedom technique, the researchers assessed participants' perceived stress, resilience, and sexual satisfaction twice. The same tools were used by the researchers to compare them and investigate any notable differences in the results.

ELIGIBILITY:
Inclusion Criteria:

* absence of any psychiatric diagnoses
* no prior exposure to courses on emotional freedom techniques
* no chronic illnesses

Exclusion Criteria:

* previously psychiatric diagnosed women
* women with previous experiences with emotional freedom techniques
* Women with chronic illness

Ages: 20 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-07-21 (Actual)

PRIMARY OUTCOMES:
Perceived Stress | 3 Months
  Perceived Stress Scale (PSS-10) which was developed by Cohen and colleagues, (1983). Perceived Stress Scale (PSS) is widely considered the gold standard instrument for measuring stress perception. This questionnaire is used to assess the degree to which a respondent finds circumstances in their life to be unpredictable, uncontrollable, and/or overwhelming. Questions on the PSS ask the respondent to rate their feelings and thoughts for the past month indicating that a relatively recent time frame is assessed. PSS designed to measure the degree to which situations in one's life are appraised as stressful. This version of the PPS had 10 items: four positive items (items 4, 5, 7, 8) and six negative items (items 1, 2, 3, 6, 9 and 10). Each item is scored on a 5-point scale, ranging from 0 (never) to 4 (very often). The positive elements' ratings are reversed, for example, 0=4, 1=3, 2=2, etc., and then summing across all 10 items, a higher score indicates more perceived stress.

SECONDARY OUTCOMES:
Resilience | 3 Months
  Connor-Davidson Resilience Scale (CD-RISC) which was developed Kathryn and Jonathan, (2003). The Connor-Davidson Resilience Scale (CD-RISC) comprises 25 items that measure resilience or capacity to change and cope with adversity. Respondents indicated their response on a 5-point Likert scale with higher scores indicating greater resilience. Scoring criteria: As for the scoring system of the CD-RISC contains 25 items, all of which carry a 5-point range of responses, as follows: not true at all (0), rarely true (1), sometimes true (2), often true (3), and true nearly all of the time (4). The scale is rated based on how the subject has felt over the past month. The total score ranges from 0-100, with higher scores reflecting greater resilience.
Sexual Satisfaction | 3 Months
  Sexual Satisfaction Index (SSI) which was developed by Leth-Nissen and colleagues, (2021). There were nine items in this edition of the SSI: five positive items (items 1, 2, 3, 8, and 9) and four negative ones (items 4, 5, 6, and 7). Every item is scored on a 5-point rating system, with the negative ratings being reversed and ranging from 1 (strongly disagree) to 5 (strongly agree). The SSI's total score falls between 1 and 45. A greater level of sexual satisfaction is indicated by a higher sum score.

CONTACTS AND LOCATIONS:
Locations (1):
- Beni-Suef University Hospital, Banī Suwayf, Beni Suweif Governorate, Egypt

REFERENCES:
- [Derived] Mohamed AF, Hamed AEM, Mohamed SSA, Othman AA, El-Tawab NAA. Effect of nursing application of emotion freedom technique on perceived stress, resilience and sexual satisfaction among women after mastectomy. BMC Nurs. 2025 Apr 15;24(1):428. doi: 10.1186/s12912-025-02977-2. PMID 40234881